CLINICAL TRIAL: NCT06299384
Title: Voice-Based AI to Scale Evaluation of Crisis Counseling in 988 Rollout
Brief Title: The Use of Voice-Based AI in 988 Crisis Counseling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lyssn.io, Inc. (Industry)
Collaborators: ProtoCall Services, Inc. (Unknown)
Responsible Party: Principal Investigator, David Atkins, Chief Executive Officer/ Research Professor, Lyssn.io, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: R44MH133517 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-03-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Suicide; Suicide and Self-harm
Keywords: Crisis Counseling; 988; Artificial Intelligence; AI
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyssn Crisis (Experimental): To compare LyssnCrisis to SAU, researchers will use a standard randomized design in which call-takers will have services-as-usual (SAU) and LyssnCrisis phases. All call-takers will start with a 4-week baseline period of SAU where LyssnCrisis is operating in the background, but does not provide AI feedback on suicide risk assessment. Lyssn team members will on-board and train the participating call-takers on the Lyssn software (i.e., reviewing calls, sharing and accessing calls for supervision), using a similar method used in the pilot field trial. After a 4-week baseline phase, call-takers will be randomly assigned to continue SAU or begin feedback with LyssnCrisis (LC) for 12 weeks.
  LC arm participants will have access to LyssnCrisis feedback tools for the duration of the 12 week period and will receive onboarding support for LyssnCrisis fidelity feedback tools.
  Interventions: Other: LyssnCrisis
- Services As Usual (No Intervention): To compare LyssnCrisis to SAU, researchers will use a standard randomized design in which call-takers will have services-as-usual (SAU) and LyssnCrisis phases. All call-takers will start with a 4-week baseline period of SAU where LyssnCrisis is operating in the background, but does not provide AI feedback on suicide risk assessment. Lyssn team members will on-board and train the participating call-takers on the Lyssn software (i.e., reviewing calls, sharing and accessing calls for supervision), using a similar method used in the pilot field trial. After a 4-week baseline phase, call-takers will be randomly assigned to continue SAU or begin feedback with LyssnCrisis (LC) for 12 weeks.
  Participants in the SAU arm will continue services-as-usual for an additional 12-week period,where participants receive ProtoCall's regular supervision and feedback. Following this period (16 total weeks of SAU), SAU arm participants will receive LyssnCrisis for 12 weeks.

INTERVENTIONS:
Other: LyssnCrisis — LyssnCrisis is an AI-based coding and feedback tool for implementation in crisis counseling settings, training counselors (call-takers) in suicide risk assessment skills.
  Arms: Lyssn Crisis

SUMMARY:
Effective training requires repeated opportunities for skills practice with performance-based feedback, which is challenging to provide at scale. This research study focuses on developing an AI-based, coding and feedback tool ("LyssnCrisis") for implementation in a nationally utilized crisis call center, training counselors (call-takers) in suicide risk assessment skills, and evaluating LyssnCrisis to improve services and client outcomes. This research study's goal is to maximize the human capacity of call-takers to help assess their callers for risk of suicidality, and thus, a core aspect of the current research is developing a novel training process that supports human call-taker capacities.

ELIGIBILITY:
Inclusion Criteria:

Must be employed at Protocall Services, Inc.

Exclusion Criteria:

Call-takers who participated in Stage 2 research will not be able to participate in Stage 3 research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Post-Call Survey | Through study completion, an average of 22 weeks.
  9 item survey utilizing LifeLine crisis call questions that measures changes in distress, perceived helpfulness, and call-taker relationship at the conclusion of a crisis call. The survey is completed by callers to ProtoCall's 988 crisis line, facilitated by the call-taker. .
Call-taker crisis counseling fidelity | Through study completion, an average of 22 weeks.
  Crisis counseling fidelity will be assessed by AI-generated scores for every recorded call, which will be analyzed via Lyssn during both SAU and LyssnCrisis phases of the study. Key fidelity metrics will include empathy, use of active listening skills, and whether the counselor asked any of the 7 key risk assessment questions (e.g., ideation, plan, past attempts).
System Usability Scale (SUS) | Through study completion, an average of 22 weeks.
  10 item survey that is a general measure of technology usability [ Rated from 1-5, 1= strongly disagree, 5 = strongly agree]
Acceptability of Intervention Measure; AIM | For Pilot: at end of 2 week LyssnCrisis period; for RCT, at end of 12-week LyssnCrisis period.
  The Acceptability of Intervention (AIM) to measure target core implementation outcomes and assess if crisis tool is acceptable, appropriate, or feasible for its stated goals. A brief, 4-item measure of a mental health professional's perception of how acceptable an innovation would be for use in their context. Each statement about the acceptability of the innovation is rated on a 5-point ordinal scale ranging from "completely disagree" to "completely agree," where higher scores indicate higher levels of acceptability.
Intervention Appropriateness Measure; IAM | Through study completion, an average of 22 weeks.For Pilot: at end of 2 week LyssnCrisis period; for RCT, at end of 12-week LyssnCrisis period.
  The Intervention Appropriateness (IAM) to measure target core implementation outcomes and assess if crisis tool is acceptable, appropriate, or feasible for its stated goals. A brief, 4-item measure of a mental health professional's perception of how appropriate an innovation would be for use in their context. Each statement about the appropriateness of the innovation is rated on a 5-point ordinal scale ranging from "completely disagree" to "completely agree," where higher scores indicate higher levels of appropriateness.
Feasibility of Intervention Measure; FIM | For Pilot: at end of 2 week LyssnCrisis period; for RCT, at end of 12-week LyssnCrisis period.
  The Feasibility of Intervention (FIM) to measure target core implementation outcomes and assess if crisis tool is acceptable, appropriate, or feasible for its stated goals. A brief, 4-item measure of a mental health professional's perception of how feasible an innovation would be for use in their context. Each statement about the feasibility of the innovation is rated on a 5-point ordinal scale ranging from "completely disagree" to "completely agree," where higher scores indicate higher levels of feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: David C Atkins, PhD, Principal Investigator — Lyssn.io, Inc.
Locations (1):
- ProtoCall Services, Inc., Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
The data collected during the development and evaluation of LyssnCrisis will be critical in refining the technology and improving crisis counseling fidelity algorithms and software design. Thus, Lyssn considers this proprietary and does not plan to share this data outside of Lyssn.io and ProtoCall based colleagues. However, dissemination of findings from this research and development effort can be accomplished through publications and presentations; researchers are targeting conferences such as the Ubiquitous Computing (UbiComp) and Computer Human Interaction (CHI) and journals such as Crisis, Implementation Science, and Journal of Consulting and Clinical Psychology.